CLINICAL TRIAL: NCT02751060
Title: Evaluation of Plasma Non-coding RNAs (miRNA-320a) as Biomarkers of Diagnosis, Prognosis and Treatment Effects in Coronary Heart Disease
Brief Title: Evaluation of Plasma Non-coding RNAs as Biomarkers in Coronary Heart Disease
Status: Enrolling by invitation | Type: Observational
Sponsor: Tongji Hospital (Other)
Responsible Party: Principal Investigator, Dao Wen Wang, Prof., Tongji Hospital
Other Study IDs: TJ-IRB20160305
Record Dates: First submitted 2016-04-20; First posted 2016-04-26 (Estimated); Last update posted 2024-04-10 (Actual); Status verified 2024-04

CONDITIONS: Coronary Disease
MeSH Terms: conditions — Coronary Disease

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 2 Years

GROUPS / COHORTS (1):
- patients with coronary heart disease symptoms
  Interventions: Other: No intervention

INTERVENTIONS:
Other: No intervention

SUMMARY:
The purpose of this study is to determine whether the expression level of miR-320a are effective as biomarker in evaluating the diagnosis, prognosis and treatment effects of coronary heart disease.

ELIGIBILITY:
Inclusion Criteria:

1. 18 years of age or older;
2. the most recent symptoms of coronary heart disease within 7 days;
3. meet one of the following conditions: A. clinical history of typical ischemic chest pain (more than 5 minutes of persistent chest pain); B. serum cardiac biomarkers positive (TnT/I or creatine kinase peak greater than 99% of URL); C. Electrocardiogram changes of myocardial ischemia.

Exclusion Criteria:

1. pregnant women or plan to;
2. participate in any drug clinical trials within 3 months;
3. patients with life-threatening complications, or the researchers determined that the survival time of patients with no more than 1 years;
4. serious neurological disease (Alzheimer's disease, Parkinson syndrome, progressive lower limbs or deaf patients);
5. previous history of cancer or tumor, or pathological examination confirmed precancerous lesions (such as breast ductal carcinoma in situ, or atypical hyperplasia of the cervix);
6. patients refused to comply with the requirements of this study to complete the research work;
7. according to the researchers, patients can not complete the study or not to comply with the requirements of this study (because of the reasons for the management or other reasons).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: 4000 outpatients or hospitalized patients with coronary heart diseasewill be enrolled in this study.
Sampling Method: Non-Probability Sample
Enrollment: 4000 (Estimated)
Dates: Start 2016-04 (Actual); Primary Completion 2025-12 (Estimated); Study Completion 2026-12 (Estimated)

PRIMARY OUTCOMES:
the plasma expression of miR-320a in coronary heart disease patients compared to control patients | up to 24 months

SECONDARY OUTCOMES:
number of participants with cardiovascular causes of death | up to 24 months
number of participants with non fatal myocardial infarction or stroke | up to 24 months
number of participants with re-hospitalization due to cardiovascular causes | up to 24 months
number of participants with all causes of mortality | up to 24 months
number of participants with myocardial infarction re-exacerbation or re-hospitalization | up to 24 months

CONTACTS AND LOCATIONS:
Overall Officials: Dao Wen Wang, Doctor, Principal Investigator — Tongji Hospital
Locations (1):
- Tongji Hospital, Wuhan, Hubei, China